CLINICAL TRIAL: NCT04123067
Title: Pioglitazone Treatment for Hyperglycemic Acute Ischemic Stroke: Effects on the Stress-Immune Response
Brief Title: Pioglitazone Treatment for Hyperglycemic Acute Ischemic Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Temporarily suspended due to Pandemic.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00011042
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Acute; Hyperglycemia; Diabetes
MeSH Terms: conditions — Stroke; Hyperglycemia; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pioglitazone treatment group (Experimental): oral administration of 45mg Pioglitazone daily for three subsequent days, initiated within 12h of stroke symptom onset
  Interventions: Drug: Pioglitazone 45 mg
- Placebo group (Placebo Comparator): Oral administration of placebo daily for three subsequent days, initiated within 12h of stroke symptom onset
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pioglitazone 45 mg — 45mg Pioglitazone daily for three subsequent days, initiated within 12h of stroke symptom onset
  Arms: Pioglitazone treatment group
Drug: Placebo oral tablet — placebo daily for three subsequent days, initiated within 12h of stroke symptom onset
  Arms: Placebo group

SUMMARY:
Study objective is to determine whether Pioglitazone (PGZ) can improve clinical outcomes in hyperglycemic acute ischemic stroke (IS). The rationale for the proposed research is to develop an acute intervention that can improve neurological recovery and decrease mortality and morbidity in high-risk diabetic stroke patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blinded stroke intervention study. Patients presenting with hyperglycemia (blood glucose level = or > than 150mg/dl) and acute stroke symptoms within 12h of onset will be randomized to either treatment with PGZ or placebo. Patients will receive oral drug vs placebo once daily for three consecutive days. Blood samples will be obtained at baseline and during the subsequent three days to collect various biomarkers of the stress-immune response following ischemic stroke. Clinical outcomes (NIH-SS and mRS) will be determined at 3 months. Secondary outcome measures are changes in the various blood biomarkers comparing both study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke Patients ages 21 and over
2. Blood sugar ≥ 150 mg/dl
3. Study drug treatment should be initiated within 12 hours after time of symptom onset, if known, or the time last known normal (if time to symptom onset is unknown)
4. MRI or CT proven ischemic stroke
5. Initial NIH SS of ≥ 2
6. Willing and able to provide consent

Exclusion Criteria:

1. Known hypersensitivity to PGZ.
2. Infection at the time of presentation as defined by body temperature > 38 degrees C , pneumonia evident on chest X-ray, urinary tract infection (positive tests for nitrites, leukocyte esterase, and bacteria on urine analysis), other acute infection per history or current use of antibiotic or antiviral treatment.
3. Active malignancy and / or autoimmune disease requiring treatment.
4. Use of immunomodulatory drugs or chemotherapy.
5. History of stroke or brain injury within the last 90 days prior to presentation.
6. Acute illness within the last 30 days which could have affected the white blood cell count.
7. Known history of clinically significant hypoglycemia.
8. Patients already taking PGZ.
9. Active liver disease (ALT and /or AST 2.5 times the upper limit of normal, total bilirubin > 1.2 mg/dl).
10. Acute decompensated heart failure, and/or admission for an acute coronary syndrome, myocardial infarction (MI), cardiac arrest, coronary artery surgery within the past 3 months and patients with New York Heart association Class III and IV heart failure.
11. History of bladder cancer
12. Pregnant and nursing women.
13. Currently incarcerated patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Bettermann, MD, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone Treatment Group | Placebo Group
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Pioglitazone Group contains 0 participants because the Responsible Party terminated the study following the enrollment of first study subject
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 72 (0) | 72 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Neurological Status
Description: NIH-Stroke scale (0-42) to assess neurological function with 0 being no deficits and 42 being the worst score
Time Frame: 90 days post stroke
Population: Subject that received Placebo was lost to follow up and 90 day outcome data was not collected.
Arm/Group | Pioglitazone Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Degree of Disability or Dependence in the Daily Activities
Description: Measured using the modified Rankin Scale (0-6) to assess neurological function with a score of 0 for no neurological deficits and a maximum of 6 for an expired patient
Time Frame: 90 days post stroke
Population: Subject that received Placebo was lost to follow up and 90 day outcome data was not collected.
Arm/Group | Pioglitazone Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Concentration of Markers of Neutrophil Activation and Function
Description: measured in blood by flow cytometry
Time Frame: 24 hours, 48 hours, and 90 days post-stroke
Population: Subject that received Placebo was lost to follow up and data was not collected for any time point
Arm/Group | Pioglitazone Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Concentration of Stress Response Markers Including Cortisol, Norepinephrine and Epinephrine
Description: measured in blood
Time Frame: 24 hours, 48 hours, and 90 days poststroke
Population: Subject that received Placebo was lost to follow up and data was not collected for any time point.
Arm/Group | Pioglitazone Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Description: Placebo Group contains 0 participants because the Responsible Party terminated the study following the enrollment of first study subject, therefore, no serious adverse events, All-cause mortality or other (Not Including Serious) Adverse Events are recorded for the placebo group.
Arm/Group | Pioglitazone Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of funding and Responsible Party relocating to another institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04123067/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04123067/ICF_001.pdf